CLINICAL TRIAL: NCT01328756
Title: A Phase 4, Open-Label, Multicentre, Safety Study of Lisdexamfetamine Dimesylate in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Lisdexamfetamine Dimesylate 2-year Safety Study in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPD489-404; 2010-020951-30 (EudraCT Number); NCT01413165 (obsolete NCT alias)
Record Dates: First submitted 2011-03-29; First posted 2011-04-05 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

ARMS (1):
- Lisdexamfetamine Dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — Optimized dose of either 30, 50 or 70 mg capsule administered once daily for 2 years
  Other Names: Vyvanse, SPD489, LDX

SUMMARY:
While the Lisdexamfetamine Dimesylate (SPD489) clinical program has studied the efficacy, safety, and tolerability of SPD489 in treating core symptoms of ADHD in children and adolescents aged 6-17 years and adults aged 18-55 years, the majority of these studies have been of short duration - up to 8 weeks.

A number of long-term studies have been undertaken (up to 1 year) and these have confirmed the safety and ongoing efficacy in this patient population.

In order to run a study with investigational medication within Poland the study changed to a Phase 3 rather than a Phase 4 study in that country. Please note that the study number remains as SPD489-404.

Study SPD489-404 has been designed to further evaluate the long-term effects of SPD489 in children and adolescents over a 2-year treatment period.

ELIGIBILITY:
Inclusion Criteria:

For subjects who participated in another SPD489 study (SPD489-317, SPD489-325, or SPD489 326):

* Subject is a male or female aged 6-17 years.
* Subject participated in SPD489-317, completed 9 weeks of treatment, and completed the 1 week post-treatment safety follow-up visit.

For subjects who have not participated in another SPD489 study:

* Subject is a male or female aged 6-17 years.
* Subject must meet DSM-IV-TR criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation.

For all subjects:

* Subject has a Baseline ADHD-RS-IV total score greater than or equal to 28.
* Subject, who is female of childbearing potential (FOCP), must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test, and a negative urine pregnancy test at Baseline, be non-lactating and agree to comply with any applicable contraceptive requirements of the protocol.
* Subject and parent/LAR are willing and able to comply with all the testing and requirements defined, including oversight of morning dosing. Specifically, the parent/LAR must be available upon awakening, at approximately 7:00 AM, to dispense the dose of Investigational Product for the duration of the study.
* Subject aged greater than or equal to 18 years has a systolic blood pressure less than or equal to 139 mmHg and a diastolic blood pressure less than or equal to 89 mmHg.
* Subject is able to swallow a capsule.

Exclusion Criteria:

For subjects who participated in another SPD489 study (SPD489-317, SPD489-325, or SPD489 326):

* Subject was terminated from a previous SPD489 study (SPD489-325 or SPD489 326) for protocol non-adherence and/or subject non-compliance and/or experienced a medication-related SAE or AE resulting in termination from the previous study.
* Subject experienced any clinically significant AEs in a prior SPD489 study (SPD489 317, SPD489-325, or SPD489-326) that, in the opinion of the Investigator, would preclude further exposure to SPD489.

For all subjects:

* Subject's symptoms are well-controlled on their currently prescribed ADHD medication with acceptable tolerability.
* Subject has a positive urine drug result at Screening.
* Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any severe comorbid Axis II disorder or severe Axis I disorder (such as Post Traumatic Stress Disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder) or other symptomatic manifestations, such as agitated states, marked anxiety, or tension.
* Subject has taken another Investigational Product or taken part in a clinical study with the exception of a prior SPD489 study (SPD489-317, SPD489 325, or SPD489 326) within 30 days prior to Screening.
* Subject weighs less than 22.7 kg (50 lbs).
* Subject is significantly overweight.
* Subject has a conduct disorder. Oppositional defiant disorder is not exclusionary.
* Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject.
* Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator
* Subject has glaucoma.
* Subject has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone (TSH) and thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Subject has any clinically significant ECG abnormality.
* Subject has any clinically significant laboratory abnormalities.
* Subject has a documented allergy, hypersensitivity, or intolerance to any active ingredient or excipients in SPD489.
* Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria.
* Subject has a history of seizures (other than infantile febrile seizures), a chronic or current tic disorder, a current diagnosis of Tourette's Disorder, or a known family history of Tourette's Disorder. Subject has a history of tics that is judged by the Investigator to be exclusionary.
* Subject has a known history of symptomatic cardiovascular or cerebrovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subject has a medical condition, other than ADHD, that requires treatment with medications that have central nervous system effects and/or affect performance. Stable use of anticholinergic or theophylline bronchodilators is not exclusionary.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2011-07-07 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (35):
- Belgium (2):
  - ZNA Antwerpen, Commandant Weynsstraat 165 Campus Hoge Beuken, Hoboken, Antwerp
  - Afdeling Psychiatrie, Leuven
- Germany (7):
  - Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim, Baden-Wurttemberg
  - Schwerpunktpraxis für Entwicklung und Lernen, Bamberg, Bavaria
  - Medizinisches Studienzentrum Würzburg, Würzburg, Bavaria
  - Praxis Dr.Christian Wolff, Hagen, North Rhine-Westphalia
  - Universitätsmedizin Berlin, Berlin
  - Praxis Dr. med. Friedrich Kaiser und Dr. med. Ingrid Marinesse, Hamburg
- Hungary (4):
  - Gyermek es Ifjusagpszichiatriai Szakrendeles es Gondozo Veress E. u. 2., Pécs, Baranya
  - Szegedi Tudomanyegyetem, Gyermek- es Ifjusagpszichiatriai Osztaly Boldogasszony sgt. 15, Szeged, Csongrád megye
  - Vadaskert Korhaz es Szakambulancia, Gyermek es Ifjusagpszichiatria Huvosvolgyi ut 116, Budapest
  - Pandy Kalman Korhaz, Gyermekpszichiatria Semmelweis u.1., Gyula
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
- Academisch Ziekenhuis Maastricht, Heerlen, Limburg, Netherlands
- Poland (3):
  - Szpital Uniwersytecki im. dr. Antoniego Jurasza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Osrodek Lecznictwa Psychiatrycznego W Toruniu, Torun, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw, Masovian Voivodeship
- Romania (3):
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu", Timișoara, Timiș County
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Bucharest
  - Spitalul Clinic de Psihiatrie Socola, Iași
- Spain (8):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Sant Joan de Deu, Servicio de Psiquiatria Infantil Passeig Sant Joan de Deu, 2 Esplugues de Llobregat, Esplugues de Llobregat, Barcelona
  - Mutua de Terrassa, Centro de Salud Mental Cap Rambla Psiquiatria Infantil Placa Doctor Robert, 5, Terrassa, Barcelona
  - Hospital Maritimo de Torremolinos, Torremolinos, Malaga
  - Clinica Universitaria de Navarra, Unidad de Psiquiatría Infantil y Adolescente, Dept. de Psiquiatria y Psicologia Medica Avenida Pio XII 36 Apartado 4209 Pamplona, Pamplona, Navarre
  - Hospital Univeritario de Canarias, Consultas Externas de Psiquiatria Ofra l La Cuesta s/n San Cristobal de la Laguna Laguna Santa Cruz, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Hospital Clinic I Provincial de Barcelona, Barcelona
- Sweden (3):
  - Child Neuropsychiatry Centre The Queen Silvia Children's Hospita Otterhallegatan 12A, Gothenburg
  - Barn och Ungdomsmedicin klinik Molnlycke Ekdalavagen 2 Box 9, Mölnlycke
  - Paediatric Neurology Children's Hospital in Huddinge, Stockholm
- United Kingdom (2):
  - Thurrock Hospital, Grays, England
  - University of Dundee, Centre for Child Health 19 Dudhope Terrace Scotland, Dundee, Scotland

REFERENCES:
- [Derived] Banaschewski T, Johnson M, Nagy P, Otero IH, Soutullo CA, Yan B, Zuddas A, Coghill DR. Growth and Puberty in a 2-Year Open-Label Study of Lisdexamfetamine Dimesylate in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2018 May;32(5):455-467. doi: 10.1007/s40263-018-0514-8. PMID 29790103
- [Derived] Coghill DR, Banaschewski T, Bliss C, Robertson B, Zuddas A. Cognitive Function of Children and Adolescents with Attention-Deficit/Hyperactivity Disorder in a 2-Year Open-Label Study of Lisdexamfetamine Dimesylate. CNS Drugs. 2018 Jan;32(1):85-95. doi: 10.1007/s40263-017-0487-z. PMID 29383572
- [Derived] Coghill DR, Banaschewski T, Nagy P, Otero IH, Soutullo C, Yan B, Caballero B, Zuddas A. Long-Term Safety and Efficacy of Lisdexamfetamine Dimesylate in Children and Adolescents with ADHD: A Phase IV, 2-Year, Open-Label Study in Europe. CNS Drugs. 2017 Jul;31(7):625-638. doi: 10.1007/s40263-017-0443-y. PMID 28667569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants from 3 antecedent studies (SPD489-317 [NCT01106430], SPD489-325 [NCT00763971], and SPD489-326 [NCT00784654]), or directly enrolled.
Pre-assignment Details: If participants from previous SDP489 studies had a gap of more than 7 days before participation in this study, they were required to have baseline Attention-Deficit/Hyperactivity Disorder (ADHD) total score of at least 28, to be enrolled. Of 348 participants screened, 314 participants were enrolled and treated.
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine dimesylate (SPD489) 30, 50 and 70 milligram (mg) capsules once daily orally during the 4-week dose optimization period and the 100-week maintenance period. At optimization period, participants started SPD489 30 mg and dose was titrated until acceptable response (30% reduction from baseline in ADHD Rating Scale-IV total score, clinical global impression-improvement [CGI-I]score of 1 or 2 with tolerable side effects) was achieved. Maximum dose was 70mg. Dose adjustments were done in dose maintenance period.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate
Started | 314
Completed | 191
Not Completed | 123
Not completed — Protocol Violation | 4
Not completed — Adverse Event | 39
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 41
Not completed — Lost to Follow-up | 5
Not completed — Other | 29

BASELINE CHARACTERISTICS:
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine dimesylate (SPD489) 30, 50 and 70 mg capsules once daily orally during the 4-week dose optimization period and the 100-week maintenance period.
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 250
Clinical Global Impressions - Severity of Illness (CGI-S) Rating [Count of Participants; unit: Participants] — The Clinical Global Impressions (CGI) Scale permits a global evaluation of the participant's severity and improvement over time. This assessment will help guide the clinician on dosing adjustments. The CGI has been used extensively in clinical studies of ADHD. CGI-S was a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants), evaluated by the Investigator.
  Participants
    Normal, not all ill | 0
    Borderline mentally ill | 0
    Mildly ill | 1
    Moderately ill | 69
    Markedly ill | 152
    Severely ill | 81
    Among the most extremely ill participants | 11
Body Weight [Mean (Standard Deviation); unit: kilogram(s)] | 46.13 (16.434)
Height [Mean (Standard Deviation); unit: centimeters] | 152.29 (16.633)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] — BMI was calculated as (weight [kilogram] per height [square meter]) at screening.
  kilogram per square meter | 19.22 (3.389)
Attention-Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV): Total Score [Mean (Standard Deviation); unit: scores on a scale] — ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria, completed by the Investigator. Each item was scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items were grouped into 2 sub-scales: hyperactivity/impulsivity (even number items 2-18 with score range of 0 to 27) and inattention (odd number items 1-17 with score range of 0 to 27). Higher scores depicted worse symptoms.
  scores on a scale | 41.1 (7.03)
ADHD-RS-IV: Inattention Subscale Score [Mean (Standard Deviation); unit: scores on a scale] — ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on DSM-IV-TR criteria, completed by the Investigator. Each item was scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items were grouped into 2 sub-scales: hyperactivity/impulsivity and inattention. Inattention subscale score consisted of odd number items 1-17 with scores ranging from 0 to 27. Higher score indicated worse symptom.
  scores on a scale | 22.1 (3.52)
ADHD-RS-IV: Hyperactivity/Impulsivity Subscore [Mean (Standard Deviation); unit: scores on a scale] — ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on DSM-IV-TR criteria, completed by the Investigator. Each item was scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items were grouped into 2 sub-scales: hyperactivity/impulsivity and inattention. Hyperactivity/impulsivity subscale score consisted of even number items 2-18 with scores ranging from 0 to 27. Higher score indicated worse symptom.
  scores on a scale | 19 (5.86)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. It included both serious and non-serious adverse event. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs were defined as treatment-emergent if they started or worsened during the period between the day of a participant's first dose of investigational product in this study and the 3 days following cessation of treatment.
Time Frame: Baseline up to 3 days after the last dose of study treatment (up to 2 years)
Population: Safety population included all participants who took at least 1 dose of Lisdexamfetamine dimesylate during this study.
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 314
participants
  Any TEAE | 282
  Serious TEAE | 28

2. Primary Outcome: Change From Baseline in Pulse Rate at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
beats per minute | 7 (11.6)

3. Primary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
mmHg | 3.2 (9.05)

4. Primary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
mmHg | 3.4 (10.33)

5. Primary Outcome: Change From Baseline in Body Weight at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: kilogram(s)
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
kilogram(s) | 2.1 (5.83)

6. Primary Outcome: Change From Baseline in Height at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: centimeter(s)
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 301
centimeter(s) | 6.1 (4.9)

7. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Last On-treatment Assessment (LOTA)
Description: BMI was calculated as (weight [kilogram] per height [square meter]).
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: kilogram per square meter
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
kilogram per square meter | -0.5 (1.72)

8. Primary Outcome: Change From Baseline in Heart Rate at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 303
beats per minute | 7.1 (13.51)

9. Primary Outcome: Change From Baseline in QT Interval at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 302
milliseconds | -10.3 (23.53)

10. Primary Outcome: Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF) at Last On-treatment Assessment (LOTA)
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 302
milliseconds | -0.6 (15.24)

11. Primary Outcome: Change From Baseline in Brief Psychiatric Rating Scale for Children (BPRSC) Total Scores at Last On-treatment Assessment (LOTA)
Description: The BPRS-C that was designed to provide a characterization of the child and adolescent psychopathology, was used to monitor participant's safety. The BPRS-C assessed 7 independent factors (3 items each), for a total of 21 items that represented behavioural disorders, depression, thinking disturbance, psychomotor excitation, withdrawal retardation, anxiety, and organicity. Each item was rated using a 7-point scale including 0 (not present), 1 (very mild), 2 (mild), 3 (moderate), 4 (moderately severe), 5 (severe), and 6 (extremely severe). Total score is the sum of each item score; range from 0 to 126. Higher score indicated worse psychology.
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Safety population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 313
scores on a scale | -10.3 (9.64)

12. Secondary Outcome: Change From Baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Total Score at Last On-treatment Assessment (LOTA)
Description: ADHD-RS-IV consisted of 18 items designed to reflect current symptomatology of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria, completed by the Investigator. Each item was scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items were grouped into 2 sub-scales: hyperactivity/impulsivity (even number items 2-18 with score range of 0 to 27) and inattention (odd number items 1-17 with score range of 0 to 27). Higher scores depicted worse symptoms.
Time Frame: Baseline (Week 0), LOTA (Week 104)
Population: Full Analysis Set (FAS) population included all participants who took at least 1 dose of SPD489 and had at least 1 on-treatment post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 299
Scores on a scale | -25.8 (11.1)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate; Change from baseline to LOTA value was assessed for differences from zero using a 2-sided, 1 sample t-test at a 0.05 significance level; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Number of Participants With Clinical Global Impression-Global Improvement (CGI-I) at Last On-treatment Assessment (LOTA)
Description: The Clinical Global Impressions (CGI) Scale permits a global evaluation of the participants' severity and improvement over time. This assessment will help guide the clinician on dosing adjustments. The CGI has been used extensively in clinical studies of ADHD. CGI-I was a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), evaluated by the Investigator.
Time Frame: LOTA (Week 104)
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 299
participants
  Very much improved | 141
  Much improved | 92
  Minimally improved | 28
  No change | 20
  Minimally worse | 13
  Much worse | 5
  Very much worse | 0

14. Secondary Outcome: Number of Participants With Clinical Global Impression-Severity of Illness (CGI-S) at Last On-treatment Assessment (LOTA)
Description: The Clinical Global Impressions (CGI) Scale permits a global evaluation of the participants' severity and improvement over time. This assessment will help guide the clinician on dosing adjustments. The CGI has been used extensively in clinical studies of ADHD. CGI-S was a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants), evaluated by the Investigator.
Time Frame: LOTA (Week 104)
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate
Number analyzed (Participants) | 299
participants
  Normal, not all ill | 73
  Borderline mentally ill | 97
  Mildly ill | 67
  Moderately ill | 39
  Markedly ill | 17
  Severely ill | 4
  Among the most extremely ill participants | 2

ADVERSE EVENTS:
Time Frame: Baseline up to 3 days after the last dose of study treatment (up to 2 years)
Description: AEs were defined as treatment-emergent if they started or worsened during the period between the day of a participant's first dose of investigational product in this study and the 3 days following cessation of treatment.
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine dimesylate (Vyvanse, SPD489) 30 to 70 mg capsule once daily orally.
Arm/Group | Lisdexamfetamine Dimesylate
Serious Adverse Events (participants affected / at risk) | 28/314
Other Adverse Events (participants affected / at risk) | 250/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (N=314)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Disbacteriosis (Gastrointestinal disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1)
Infectious peritonitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Mumps (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2)
Retroperitoneal abscess (Infections and infestations) | 1 (1)
Agitation postoperative (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 6 (7)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (N=314)
Abdominal pain (Gastrointestinal disorders) | 29 (37)
Abdominal pain upper (Gastrointestinal disorders) | 28 (34)
Nausea (Gastrointestinal disorders) | 31 (41)
Vomiting (Gastrointestinal disorders) | 27 (33)
Irritability (General disorders) | 36 (39)
Pyrexia (General disorders) | 31 (40)
Gastroenteritis (Infections and infestations) | 18 (21)
Nasopharyngitis (Infections and infestations) | 73 (129)
Pharyngitis (Infections and infestations) | 16 (18)
Weight decreased (Investigations) | 63 (68)
Decreased appetite (Metabolism and nutrition disorders) | 170 (214)
Headache (Nervous system disorders) | 68 (139)
Depressed mood (Psychiatric disorders) | 19 (20)
Initial insomnia (Psychiatric disorders) | 38 (46)
Insomnia (Psychiatric disorders) | 60 (75)
Tic (Psychiatric disorders) | 18 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (25)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (24)

LIMITATIONS AND CAVEATS:
Since this study is an open-label trial, results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.